CLINICAL TRIAL: NCT04871672
Title: Effects of Pilates Exercises on Core Stability After Recovery From COVID -19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Wafaa Mahmoud Amin, Wafaa Mahmoud Amin, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sponsor-Investigator:
Record Dates: First submitted 2021-04-24; First posted 2021-05-04 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Covid19; Pilates, Core Stability
MeSH Terms: conditions — COVID-19 | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to two groups:
  1. pilates and home exercises (PAH) group
  2. home exercises group (COH)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pilates and home exercises (PAH) group (Experimental): these subjects will receive pilates and home exercises.
  Interventions: Other: Pilates Exercises; Other: Home Exercise program
- control home exercises group (COH) (Active Comparator): these subjects will receive only home exercises.
  Interventions: Other: Home Exercise program

INTERVENTIONS:
Other: Pilates Exercises — basic five pilates intermediate workout based on the principles of Pilates
  Arms: pilates and home exercises (PAH) group
Other: Home Exercise program — home exercise

SUMMARY:
This study will be conducted in the Department of physical therapy, College of Applied Medical Sciences,Jazan University, to Effects of Pilates Exercises on core stability after Recovery from COVID - 19

DETAILED DESCRIPTION:
145 male and female students who had infected with covid 19 with age 19 to 26 years old, will be recruited from the College of Applied Medical Sciences, Jazan University. Subjects will be randomly assigned to a pilates and home exercises (PAH) group or a control group who will perform only home exercises (COH)

Four core endurance tests will be performed to assess the core stability

Pilates exercise program will be composed of Pilates mat exercise program for a period of 12 weeks and three sessions every week.

Each session took one hour. Every session started with 10 minutes of simple stretching movements to warm-up followed by the main part of the exercise plan for 40 min, followed by 10 minutes, some cool-down stretching.

When the 12-week study period will over, the core stability will be assessed by the endurance tests and Prokin system for balance

ELIGIBILITY:
Inclusion Criteria:

1. Persons who had mild to moderate covid- 19 illness.
2. Asymptomatic period of at least seven days (without chest pain, breathlessness).
3. No musculoskeletal damage.
4. No pregnancy.
5. No visually identified asymmetries in the spinal trunk and lower limbs.
6. None of the subjects has a history of balance training
7. Subjects will not have any diseases of the central nervous system.
8. Subjects with body mass index (BMI)<25 kg/m2.

Exclusion Criteria:

1. Persons who had more severe covid 19 illnesses and were hospitalized.
2. Persons who had during their illness chest pain breathlessness, palpitation, symptoms, and signs of heart failure.

9. Subjects with cardiopulmonary disorders. 3. A history of previous back or abdominal surgery/injury 4. Evidence of a systemic or musculoskeletal disease within the past six months

-

Ages: 19 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2021-12-26 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of core stability: endurance capacity of anterior deep trunk muscles | at the date of the first session and at the last session after 12 weeks
  Abdominal fatigue test: is an isometric trunk flexor test
Evaluation of core stability: assesses the functioning of trunk extensor muscles | at the date of the first session and at the last session after 12 weeks
  Sorensen back-extension endurance
Evaluation of core stability: Prone Plank test | at the date of the first session and at the last session after 12 weeks
  Prone Plank test
Evaluation of core stability: Endurance capacity of lateral core muscles particularly the quadrates lumborum | at the date of the first session and at the last session after 12 weeks
  Side Plank Tests
Evaluation of core stability: balance test by Prokin system for perimeter parameter with opened eyes, measured in mm | 30 seconds
  Eyes Open perimeter (EOPM), measured in mm
Evaluation of core stability: balance test by Prokin system for perimeter parameter with closed eyes, measured in mm | 30 seconds
  Eyes closed perimeter (ECPM), measured in mm
Evaluation of core stability: balance test by Prokin system for ellipse area parameter with Opened eyes, measured in mm | 30 seconds
  Eyes Open ellipse area (EOEA) measured in mm2
Evaluation of core stability: balance test by Prokin system for ellipse area parameter with closed eyes, measured in mm | 30 seconds
  Eyes closed ellipse area (ECEA) measured in mm2

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan University, Riyadh, Jazan Region, Saudi Arabia